CLINICAL TRIAL: NCT05623189
Title: A Phase 2b, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of HTD1801 in Adult Subjects With Nonalcoholic Steatohepatitis (NASH) and Liver Fibrosis Who Have Type 2 Diabetes (T2DM) or Pre-Diabetes
Brief Title: HTD1801 in Adults With Nonalcoholic Steatohepatitis and Liver Fibrosis Who Have Type 2 Diabetes or Pre-Diabetes
Acronym: CENTRICITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTD1801.PCT014; The CENTRICITY Study (Other: HighTide Therapeutics)
Record Dates: First submitted 2022-10-11; First posted 2022-11-21 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Type 2 Diabetes
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This phase 2b, double-blind, placebo-controlled, multicenter study will evaluate the effect of HTD1801 on histologic improvements in adult subjects with non-alcoholic steatohepatitis (NASH) and liver fibrosis who have type 2 diabetes mellitus or pre-diabetes. Approximately 210 subjects with biopsy-confirmed NASH and evidence of stage 2 or stage 3 liver fibrosis will be randomized 2:1 to receive HTD1801 1250 mg twice daily (BID) or placebo BID. Subjects will receive investigational product for up to 60 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HTD1801 (Experimental): HTD1801,1250 mg, BID
  Interventions: Drug: HTD1801
- placebo (Placebo Comparator): placebo, BID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801,1250 mg, BID
  Other Names: HTD1801 capsules
  Arms: HTD1801
Drug: Placebo — Placebo, BID
  Other Names: placebo capsules
  Arms: placebo

SUMMARY:
A phase 2b, multicenter, randomized, double-blind, placebo-controlled study of HTD1801 in adult subjects with non-alcoholic steatohepatitis and liver fibrosis who have type 2 diabetes mellitus or pre-diabetes.

DETAILED DESCRIPTION:
This phase 2b, double-blind, randomized, placebo-controlled, multicenter study will evaluate the effect of HTD1801, 1250 mg twice daily (BID) compared to placebo BID on histologic improvements in adult subjects with non-alcoholic steatohepatitis and liver fibrosis who have type 2 diabetes mellitus or pre-diabetes.

The study will enroll approximately 210 subjects with biopsy-confirmed non-alcoholic steatohepatitis and evidence of stage 2 or stage 3 liver fibrosis. Subjects will receive investigational product for up to 60 weeks.

ELIGIBILITY:
Key Inclusion criteria:

* Clinical diagnosis of non-alcoholic steatohepatitis (NASH) upon central read of a liver biopsy obtained no more than 6 months before Day 0.
* Histologic evidence of fibrosis stage 2 or stage 3 as defined by the non-alcoholic steatohepatitis (NASH) clinical research network (CRN) scoring of fibrosis.
* Clinically documented diagnosis of type 2 diabetes mellitus for at least 6 months prior to screening or prediabetes at screening.
* BMI >25 kilograms/meters squared (>23 kilograms/meters squared if Asian).

Key Exclusion criteria:

* Fibrosis stage 4.
* History of alcohol or substance abuse or dependence.
* Liver disease unrelated to non-alcoholic steatohepatitis.
* History of significant cardiovascular disease.
* History of type 1 diabetes.
* Inability or unwillingness to undergo 2 planned liver biopsies OR 1 planned biopsy if historical liver biopsy was used to confirm eligibility at entry.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2022-12-27 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint | Up to 60 Weeks
  A decrease of ≥2-points in non-alcoholic fatty liver disease activity score (NAS) with ≥1-point decrease of either lobular inflammation or ballooning and no worsening of fibrosis; OR Resolution of non-alcoholic steatohepatitis (NASH) (defined as the overall histopathologic interpretation of 1) "no fatty liver disease" or 2) "fatty liver disease (simple or isolated steatosis) without steatohepatitis AND a non-alcoholic fatty liver disease activity score (NAS) of 0 for ballooning and 0-1 for inflammation and no worsening of fibrosis.
  Nonalcoholic fatty liver disease activity score (NAS) is a histological scoring system that assesses a liver biopsy and gives scores for steatosis (0-3), lobular inflammation (0-3), and hepatocyte ballooning (0-2). The higher the score the more severe the disease. The total range for non-alcoholic fatty liver disease activity score (NAS) is between 0 to 8. The lower the score the better the outcome.

SECONDARY OUTCOMES:
Endpoint 1 | Up to 60 Weeks
  Percentage of subjects with resolution of non-alcoholic steatohepatitis (NASH) on overall histopathological reading
Endpoint 2 | Up to 60 Weeks
  Percentage of subjects with resolution of non-alcoholic steatohepatitis hepatitis (NASH) and at least a 2-point improvement in non-alcoholic fatty liver disease (NAFLD) activity score (NAS) and no worsening of liver fibrosis
Endpoint 3 | Up to 60 Weeks
  Percentage of subjects with a ≥1-stage improvement in liver fibrosis.
Endpoint 4 | Up to 60 Weeks
  Percentage of subjects with a ≥1-stage improvement in liver fibrosis and no worsening of non-alcoholic steatohepatitis (NASH).
Endpoint 5 | Up to 60 Weeks
  Percentage of subjects with a ≥2-stage improvement in liver fibrosis.
Endpoint 6 | Up to 60 Weeks
  Percentage of subjects with a ≥2-point improvement in non-alcoholic fatty liver disease activity score (NAS) and no worsening of liver fibrosis.
Endpoint 7 | Up to 60 Weeks
  Percentage of subjects with an improvement in each of the individual non-alcoholic fatty liver disease activity score (NAS) components (ballooning, inflammation, or steatosis).
Endpoint 8 | Up to 60 Weeks
  Percentage of subjects with improvement of non-alcoholic steatohepatitis (NASH) based on overall histopathologic interpretation.
Endpoint 9 | Up to 60 Weeks
  Absolute and percent change in alanine aminotransferase (ALT) from baseline to end of treatment.
Endpoint 10 | Up to 60 Weeks.
  Absolute and percent change in aspartate aminotransferase (AST) from baseline to end of treatment.
Endpoint 11 | Up to 60 Weeks
  Absolute and percent change in gamma-glutamyl transferase (GGT) from baseline to end of treatment.
Endpoint 12 | Up to 60 Weeks
  Absolute and percent change in total bilirubin from baseline to end of treatment.
Endpoint 13 | Up to 60 Weeks
  Absolute and percent change in direct bilirubin from baseline to end of treatment.
Endpoint 14 | Up to 60 Weeks
  Absolute and percent change in hemoglobin A1c (HbA1c) from baseline to end of treatment.
Endpoint 15 | Up to 60 Weeks
  Absolute and percent change in fasting plasma glucose from baseline to end of treatment.
Endpoint 16 | Up to 60 Weeks
  Absolute and percent change in body weight from baseline to end of treatment.
Endpoint 17 | Up to 60 Weeks
  Absolute and percent change in body mass index (BMI) from baseline to end of treatment.
Endpoint 18 | Up to 60 Weeks
  Absolute and percent change in hip circumference from baseline to end of treatment.
Endpoint 19 | Up to 60 Weeks
  Absolute and percent change in waist circumference from baseline to end of treatment.
Endpoint 20 | Up to 60 Weeks
  Absolute and percent change in total cholesterol from baseline to end of treatment.
Endpoint 21 | Up to 60 Weeks
  Absolute and percent change in low-density lipoprotein cholesterol (LDL-c) from baseline to end of treatment.
Endpoint 22 | Up to 60 Weeks
  Absolute and percent change in lipoprotein A (Lpa) from baseline to end of treatment.
Endpoint 23 | Up to 60 Weeks
  Absolute and percent change in high-density lipoprotein cholesterol (HDL-c) from baseline to end of treatment.
Endpoint 24 | Up to 60 Weeks
  Absolute and percent change in triglycerides from baseline to end of treatment.
Endpoint 25 | Up to 60 Weeks
  Absolute and percent change in apolipoprotein B (ApoB) from baseline to end of treatment.
Endpoint 26 | Up to 60 Weeks
  Absolute and percent change in liver stiffness as measured by vibration-controlled transient elastography (VCTE) using FibroScan® device from baseline to end of treatment.
  The VCTE score is measured in Kilopascal Pressure Unit (kPa) and ranges from 2 to 75 kPa. The higher the kPa score the more severe the liver stiffness.
Endpoint 27 | Up to 60 Weeks
  Absolute and percent change in liver fat content as measured by controlled attenuation parameter (CAP) using FibroScan® device from baseline to end of treatment.
  The controlled attenuation parameter (CAP) score is measured in decibels per meter (dB/m) it ranges from 100 to 400 dB/m. The higher the controlled attenuation parameter (CAP) score the more severe the steatosis.
Endpoint 28 | Up to 60 Weeks
  Absolute and percent change in the FibroScan-AST (FAST) score from baseline to end of treatment.
  Fast score will be calculated based on LSM, CAP and AST values using FAST equation. An equal to or more than 0.35 value thru equal or less than 0.81 value is positive predictive value for nonalcoholic steatohepatitis and a negative predictive value from 0.73 to 1.0.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Di Bisceglie, MD, FACP, FAASLD, Study Director — Hightide Therapeutics USA, LLC
Locations (45):
- United States (43):
  - The Institute for Liver Health (Arizona Liver Health), Chandler, Arizona
  - Arizona Liver Health - Glendae, Peoria, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Aizona Liver Health, Tucson, Arizona
  - San Fernando Valley Health Institute, Canoga Park, California
  - Clinnova Research Solutions, Garden Grove, California
  - Catalina Research Institute, Montclair, California
  - California Liver Institute, Pasadena, California
  - Inland Empire Liver Foundation, Rialto, California
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Tampa Bay Medical Research, Inc., Clearwater, Florida
  - Covenant Metabolic Specialists - Fort Meyers, Fort Myers, Florida
  - Evolution Clinical Trials, Inc., Hialeah Gardens, Florida
  - ClinCloud LLC Maitland, Maitland, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Floridain Clinical Research, Miami Lakes, Florida
  - Covenant Metabolic Specialists - Sarasota, Sarasota, Florida
  - Theia Clinical Research LLC, Temple Terrace, Florida
  - ClinCloud LLC Melbourn, Viera, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Conquest Research, Winter Park, Florida
  - Louisvill Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Tandem Clinical Research, Marrero, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Jubilee Clinical Research, Inc., Las Vegas, Nevada
  - Tandem Clinical Research GI - New York, New York, New York
  - Lucas Research - Diabetes and Endocrinology, Morehead City, North Carolina
  - Clinical Research Institute of Ohio, Westlake, Ohio
  - Palmetto Clinical Research, Summerville, South Carolina
  - ClinSearch LLC, Chattanooga, Tennessee
  - Premier Research, Clarksville, Tennessee
  - Texas Clinical Research Institute, Arlington, Texas
  - Pinnacle Clinical Research, Austin, Texas
  - South Texas Research Institute, Brownsville, Texas
  - EPIC Medical Research, DeSoto, Texas
  - Pinnacle Research, Georgetown TX, Georgetown, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Pinnacle Clinical Research San Antonio, San Antonio, Texas
  - Impact Research Institute, Waco, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
  - Liver Institute NW, Seattle, Washington
- Chinese University of Hong Kong Prince of Wales Hospital, Shatin, Hong Kong
- FDI Clinical Research, San Juan, Munoz Rivera San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No